CLINICAL TRIAL: NCT05376462
Title: An Interventional Randomized Controlled Trial of the Quantra® System With the QStat® Cartridge in Trauma
Brief Title: Quantra® System With the QStat® Cartridge in Trauma
Status: Terminated | Type: Observational
Why Stopped: Only Phase 1 (observational) completed. Did not proceed to Phase 2 due to site time constraints/competing priorities.
Sponsor: HemoSonics LLC (Industry)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: HEMCS-039
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Trauma; Coagulation Defect; Bleeding
Keywords: Quantra; QStat; Viscoelastic testing
MeSH Terms: conditions — Wounds and Injuries; Hemostatic Disorders; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Quantra System with the QStat Cartridge: Viscoelastic testing using the Quantra System with the QStat Cartridge.
  Interventions: Diagnostic Test: Quantra System with the QStat Cartridge

INTERVENTIONS:
Diagnostic Test: Quantra System with the QStat Cartridge — Whole blood viscoelastic test system that provides an assessment of the patient's coagulation status.

SUMMARY:
This is a prospective, single-center, observational study to assess the Quantra QStat System in trauma patients.

DETAILED DESCRIPTION:
This is a prospective, single-center, observational study to assess the performance of the Quantra QStat System in trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years; Children under the age of 18 are protected by adults under guardianship or by court order.
* Subject is a trauma patient experiencing traumatic injuries requiring a full trauma team response according to site's level 1of trauma team activation criteria.
* Subject, or subject's legally authorized representative (LAR), is willing to provide informed consent, either prospectively or by deferred consent.

Exclusion Criteria

* Subject is pregnant.
* Subject is currently enrolled in a distinct study that might confound the result of the proposed study.
* Subject is not covered by social security.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma patients requiring a full trauma team response.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Total units of red blood cells (RBC) transfused | 24 hours post-presentation for trauma subjects
  The primary endpoint of Phase II will be the total units of red blood cells (RBC) transfused and administered 24 hours post-presentation for trauma subjects.

SECONDARY OUTCOMES:
Total number of units (cc) of platelets, fibrinogen, fresh frozen plasma and TXA transfused | 48 hours after admission to the hospital
  Total number of units (cc) of platelets, fibrinogen, fresh frozen plasma and TXA administered within at 48 hrs after admission to the hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Universitaire de Lille, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No
No plan to share individual data.